CLINICAL TRIAL: NCT00687336
Title: Phase IV Study Comparing Helicobacter Pylori Empiric Eradication With Test-Guided Treatment in Patients With Peptic Ulcer Bleeding
Brief Title: Helicobacter Pylori Empiric Treatment in Ulcer Bleeding
Acronym: HETUB
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Sabadell (Other)
Collaborators: Corporacion Parc Tauli (Other); Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government)
Responsible Party: Dr. Xavier Calvet Calvo, Hospital de Sabadell
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIR2007/058
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Last update posted 2009-07-08 (Estimated); Status verified 2009-07

CONDITIONS: Peptic Ulcer Hemorrhage
Keywords: Helicobacter pylori; Treatment; Upper gastrointestinal bleeding
MeSH Terms: conditions — Peptic Ulcer Hemorrhage; Gastrointestinal Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Empirical eradication treatment
  Interventions: Other: Empirical Hp eradication
- 2 (Active Comparator): Eradication treatment according to a diagnostic test (URT, histological test, breath test or serology).
  Interventions: Other: Eradication treatment guided by a positive test

INTERVENTIONS:
Other: Empirical Hp eradication — Empirical Helicobacter pylori treatment initiated immediately after oral intake is resumed
  Other Names: Standard Hp eradication treatment
  Arms: 1
Other: Eradication treatment guided by a positive test — Eradication treatment given if there is at least one positive diagnostic test (URT, histological test, breath test or serology) for Helicobacter pylori.
  Other Names: Standard Hp treatment
  Arms: 2

SUMMARY:
The goal of the study is to compare the effectiveness of empirical Helicobacter pylori treatment compared with treatment depending on diagnostic tests for Helicobacter pylori in patients with Upper gastrointestinal bleeding due to peptic ulcer. Main hypothesis is that empirical treatment will reduce the number of patients lost to follow-up thus improving the cure rates of Hp infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18.
* Informed Consent signed.
* Diagnosis of no variceal upper gastrointestinal bleeding secondary to a duodenal ulcer, erosive duodenitis or gastric ulcer.
* Life expectancy longer than 6 months.
* Able to attend further clinical controls.
* Absence of the following exclusion criteria.

Exclusion Criteria:

* Previous eradication treatment.
* Use of antibiotics 2 weeks prior to inclusion.
* Need for Antisecretor treatment that cannot be stopped to perform the breath test.
* Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2008-03; Primary Completion 2010-05 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Helicobacter pylori eradication rate | two years

SECONDARY OUTCOMES:
Economical evaluation through cost-effectivity study of the empiric erradicator Helicobacter pylori treatment. | two years

CONTACTS AND LOCATIONS:
Overall Officials: Pilar Garcia, Dra., Principal Investigator — Hospital de Sabadell; Xavier Calvet, Dr., Study Chair — Hospital de Sabadell
Locations (1):
- Hospital de Sabadell, Institut Universitari Parc Tauli, Sabadell, Barcelona, Spain

REFERENCES:
- [Background] Calam J. Helicobacter pylori. Eur J Clin Invest. 1994 Aug;24(8):501-10. doi: 10.1111/j.1365-2362.1994.tb01099.x. No abstract available. PMID 7982436
- [Background] Lambert JR, Lin SK, Aranda-Michel J. Helicobacter pylori. Scand J Gastroenterol Suppl. 1995;208:33-46. doi: 10.3109/00365529509107760. PMID 7777803
- [Background] Houghton J, Wang TC. Helicobacter pylori and gastric cancer: a new paradigm for inflammation-associated epithelial cancers. Gastroenterology. 2005 May;128(6):1567-78. doi: 10.1053/j.gastro.2005.03.037. PMID 15887152
- [Background] Kuipers EJ, Thijs JC, Festen HP. The prevalence of Helicobacter pylori in peptic ulcer disease. Aliment Pharmacol Ther. 1995;9 Suppl 2:59-69. PMID 8547530
- [Background] Gisbert JP, Boixeda D, Aller R, de la Serna C, Sanz E, Martin de Argila C, Abraira V, Garcia Plaza A. [Helicobacter pylori and digestive hemorrhage due to duodenal ulcer: the prevalence of the infection, the efficacy of 3 triple therapies and the role of eradication in preventing a hemorrhagic recurrence]. Med Clin (Barc). 1999 Feb 13;112(5):161-5. Spanish. PMID 10091208
- [Background] Gisbert JP, Blanco M, Mateos JM, Fernandez-Salazar L, Fernandez-Bermejo M, Cantero J, Pajares JM. H. pylori-negative duodenal ulcer prevalence and causes in 774 patients. Dig Dis Sci. 1999 Nov;44(11):2295-302. doi: 10.1023/a:1026669123593. PMID 10573377
- [Background] Soll AH, Weinstein WM, Kurata J, McCarthy D. Nonsteroidal anti-inflammatory drugs and peptic ulcer disease. Ann Intern Med. 1991 Feb 15;114(4):307-19. doi: 10.7326/0003-4819-114-4-307. PMID 1987878
- [Background] Laine L, Peterson WL. Bleeding peptic ulcer. N Engl J Med. 1994 Sep 15;331(11):717-27. doi: 10.1056/NEJM199409153311107. No abstract available. PMID 8058080
- [Background] Coghlan JG, Gilligan D, Humphries H, McKenna D, Dooley C, Sweeney E, Keane C, O'Morain C. Campylobacter pylori and recurrence of duodenal ulcers--a 12-month follow-up study. Lancet. 1987 Nov 14;2(8568):1109-11. doi: 10.1016/s0140-6736(87)91545-5. PMID 2890019
- [Background] Marshall BJ, Goodwin CS, Warren JR, Murray R, Blincow ED, Blackbourn SJ, Phillips M, Waters TE, Sanderson CR. Prospective double-blind trial of duodenal ulcer relapse after eradication of Campylobacter pylori. Lancet. 1988 Dec 24-31;2(8626-8627):1437-42. doi: 10.1016/s0140-6736(88)90929-4. PMID 2904568
- [Background] Graham DY, Hepps KS, Ramirez FC, Lew GM, Saeed ZA. Treatment of Helicobacter pylori reduces the rate of rebleeding in peptic ulcer disease. Scand J Gastroenterol. 1993 Nov;28(11):939-42. doi: 10.3109/00365529309098288. PMID 8284627
- [Background] Rokkas T, Karameris A, Mavrogeorgis A, Rallis E, Giannikos N. Eradication of Helicobacter pylori reduces the possibility of rebleeding in peptic ulcer disease. Gastrointest Endosc. 1995 Jan;41(1):1-4. doi: 10.1016/s0016-5107(95)70266-0. PMID 7698617
- [Background] Macri G, Milani S, Surrenti E, Passaleva MT, Salvadori G, Surrenti C. Eradication of Helicobacter pylori reduces the rate of duodenal ulcer rebleeding: a long-term follow-up study. Am J Gastroenterol. 1998 Jun;93(6):925-7. doi: 10.1111/j.1572-0241.1998.00278.x. PMID 9647020
- [Background] Castro-Fernandez M, Sanchez-Munoz D, Garcia-Diaz E, Miralles-Sanchiz J, Vargas-Romero J. Diagnosis of Helicobacter pylori infection in patients with bleeding ulcer disease: rapid urease test and histology. Rev Esp Enferm Dig. 2004 Jun;96(6):395-8; 398-401. doi: 10.4321/s1130-01082004000600005. English, Spanish. PMID 15230669
- [Background] Gisbert JP, Abraira V. Accuracy of Helicobacter pylori diagnostic tests in patients with bleeding peptic ulcer: a systematic review and meta-analysis. Am J Gastroenterol. 2006 Apr;101(4):848-63. doi: 10.1111/j.1572-0241.2006.00528.x. Epub 2006 Feb 22. PMID 16494583
- [Background] Gisbert JP, Calvet X, Gomollon F, Mones J; Grupo Conferencia Espanola de Consenso sobre Helicobacter pylori. [Eradication treatment of Helicobacter pylori. Recommendations of the II Spanish Consensus Conference]. Med Clin (Barc). 2005 Sep 10;125(8):301-16. doi: 10.1157/13078424. No abstract available. Spanish. PMID 16159556
- [Background] Guell M, Artigau E, Esteve V, Sanchez-Delgado J, Junquera F, Calvet X. Usefulness of a delayed test for the diagnosis of Helicobacter pylori infection in bleeding peptic ulcer. Aliment Pharmacol Ther. 2006 Jan 1;23(1):53-9. doi: 10.1111/j.1365-2036.2006.02726.x. PMID 16393280
- [Background] Garcia-Altes A, Jovell AJ, Serra-Prat M, Aymerich M. Management of Helicobacter pylori in duodenal ulcer: a cost-effectiveness analysis. Aliment Pharmacol Ther. 2000 Dec;14(12):1631-8. doi: 10.1046/j.1365-2036.2000.00871.x. PMID 11121912
- [Background] Sung JJ, Leung WK, Suen R, Leung VK, Chan FK, Ling TK, Lau JY, Lee YT, Ng EK, Cheng AF, Chung SC. One-week antibiotics versus maintenance acid suppression therapy for Helicobacter pylori-associated peptic ulcer bleeding. Dig Dis Sci. 1997 Dec;42(12):2524-8. doi: 10.1023/a:1018816729449. PMID 9440631
- [Background] Gisbert JP, Gonzalez L, de Pedro A, Valbuena M, Prieto B, Llorca I, Briz R, Khorrami S, Garcia-Gravalos R, Pajares JM. Helicobacter pylori and bleeding duodenal ulcer: prevalence of the infection and role of non-steroidal anti-inflammatory drugs. Scand J Gastroenterol. 2001 Jul;36(7):717-24. doi: 10.1080/003655201300191978. PMID 11444470
- [Background] Marshall BJ, Warren JR. Unidentified curved bacilli in the stomach of patients with gastritis and peptic ulceration. Lancet. 1984 Jun 16;1(8390):1311-5. doi: 10.1016/s0140-6736(84)91816-6. PMID 6145023
- [Background] Pellicano R, Peyre S, Leone N, Repici A, De Angelis C, Rizzi R, Rizzetto M, Ponzetto A. The effect of the eradication of Helicobacter pylori infection on hemorrhage because of duodenal ulcer. J Clin Gastroenterol. 2001 Mar;32(3):222-4. doi: 10.1097/00004836-200103000-00008. PMID 11246348